CLINICAL TRIAL: NCT00935428
Title: Causes and Circumstances of Horse Related Injuries and Impact on Quality of Life
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB e4084
Record Dates: First submitted 2009-04-15; First posted 2009-07-09 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Injury
Keywords: Equestrian injury; Horse injury; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Horse-related activity can be risky. Horses are the leading cause of animal-related fatalities in Oregon and Oregon's annual death rate from animals is 45% higher than the national rate. By interviewing injured equestrians, the investigators may be able to determine patterns of decision-making and behavior from their collective experience and develop useful safety recommendations. The investigators will also determine the impact that the injury has had on quality of life. The long-term goal of the investigators research is to develop safety and prevention recommendations and a horse-related injury prevention program to reduce the number of horse related injuries.

DETAILED DESCRIPTION:
Introduction and Background:

Horse-related activity (HRA) can be risky. The National Electronic Injury Surveillance System (NEISS) estimated that in 2006, 68,060 Americans went to a U.S. emergency room with horse-related injuries (HRI), of which 5,676 were hospitalized. However, Thomas et al estimated that 102,904 people each year from 2001 to 2003 were treated for HRI in emergency rooms nationwide. In Oregon, horses are the leading cause of animal-related fatalities in Oregon and Oregon's annual death rate from animals is 45% higher than the national rate. In a survey of 679 Northwest equestrians in Oregon, Washington, and Idaho, 81% riders reported at least one injury during their career, and 1 in 5 equestrians required hospitalization, surgery, or sustained permanent disability as a result of a HRI.

The long-term goal of our research is to develop a horse-related injury prevention program. Our preliminary study indicated that lower levels of experience were strong indicators of greater risk. The period of greatest danger appears to be during the initial 100 hours of HRA, with the incidence of injury nearly 8 times greater among novices as compared to instructors or professionals. The extent to which HRI is preventable is currently not clear, but it may be substantial. 64% of injured, experienced riders believed their incident was preventable and 47% altered their riding habits as a result.

Rationale:

There is a need to develop specific safety and prevention recommendations to reduce the number of HRIs. We intend to retrospectively determine what decisions, conditions, or other influential circumstances occurred that led to the subject's injury incident and to question the subject whether any measures could have prevented the incident from occurring. By interviewing injured equestrians, we may be able to determine patterns of decision-making and behavior from their collective experience and develop useful safety recommendations.

The investigators will also interview injured equestrians to determine the impact that the injury has had on their quality of life. There is very little information in the literature on this subject. One study indicated that in the pediatric population, 41% of injured children and adolescents had residual complaints and were still hampered in their daily activities an average of 4 years after HRI. If we can document what we suspect will be a high impact of HRI on quality of life in both adults and children, the imperative to develop injury prevention measures will be further supported.

2. Briefly summarize how participants are recruited.

The Trauma Service at OHSU keeps a state-mandated registry of all patients admitted to the Trauma Service that can be searched by injury diagnosis code. Demographic, injury, and hospital outcome data can be easily obtained and matched. Consenting subjects who were treated at OHSU between January 1, 2001 and September 20, 2008 will be contacted by mail and asked to participate in this study. Potential subjects who are currently > 18 years of age can be included in the study if a Child Assent Form has been completed and a legally authorized representative (LAR) provides consent for study participation. . Investigators will be available to answer any questions that subjects may have concerning the study.

3. Briefly describe the procedures subjects will undergo.

This study involves responding to an electronic survey that will be emailed to subjects agreeing to participate in this research study. Subjects will not undergo any physical procedures. The researchers may contact study participants by email or telephone if necessary, to clarify responses from the survey questionnaire.

4. If applicable, briefly describe survey/interview instruments used.

Study participants will respond to an equestrian survey that asks questions about the horse-related injury, including causes and circumstances surrounding the injury, experience and skill level at the time of injury, safety equipment used, ideas on how the injury might have been prevented, how it has impacted quality of life, and current health status, work status, and activity level. Study participants will also complete the Rand 36-Item Health Survey, a short survey that evaluates health status. A single survey, emailed to the subject, will include both the equestrian survey and the Rand 36. Completion of the survey will require approximately 30 minutes.

5. Briefly describe how the data will be analyzed to address the purpose of the protocol.

The responses to our study questionnaires will allow us to perform statistical analysis to determine the causes and circumstances surrounding the injury to see if safety prevention measures can be identified. It will also assess the impact of the injury on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been treated at OHSU from January 1, 2001 through September 30, 2008 for any horse related traumatic injury.
* The subject will have signed an IRB approved written informed consent and HIPAA authorization to participate in the study.
* Subjects must have access to the internet and an e-mail account to participate in the survey.
* Subjects must be able to complete surveys written in English.

Exclusion Criteria:

* Subjects who are deceased.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be identified through the OHSU Trauma Registry. Patients who were treated from January 1, 2001 through September 30, 2008 for any horse related injury will be invited to participate in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Mayberry, MD, FACS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Thomas KE, Annest JL, Gilchrist J, Bixby-Hammett DM. Non-fatal horse related injuries treated in emergency departments in the United States, 2001-2003. Br J Sports Med. 2006 Jul;40(7):619-26. doi: 10.1136/bjsm.2006.025858. Epub 2006 Apr 12. PMID 16611723
- [Background] Mayberry JC, Pearson TE, Wiger KJ, Diggs BS, Mullins RJ. Equestrian injury prevention efforts need more attention to novice riders. J Trauma. 2007 Mar;62(3):735-9. doi: 10.1097/ta.0b013e318031b5d4. PMID 17414356
- [Background] Ball CG, Ball JE, Kirkpatrick AW, Mulloy RH. Equestrian injuries: incidence, injury patterns, and risk factors for 10 years of major traumatic injuries. Am J Surg. 2007 May;193(5):636-40. doi: 10.1016/j.amjsurg.2007.01.016. PMID 17434372
- [Background] Dekker R, Van Der Sluis CK, Kootstra J, Groothoff JW, Eisma WH, Duis HJ. Long-term outcome of equestrian injuries in children. Disabil Rehabil. 2004 Jan 21;26(2):91-6. doi: 10.1080/09638280310001629688. PMID 14668145
- [Result] Guyton K, Houchen-Wise E, Peck E, Mayberry J. Equestrian injury is costly, disabling, and frequently preventable: the imperative for improved safety awareness. Am Surg. 2013 Jan;79(1):76-83. PMID 23317616

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective review of patients with horse-related injuries evaluated at OHSU Hospital from 2001 - 2008
Groups:
- Patients Injured: Those patients evaluated at OHSU Hospital with horse related injuries
Period: Overall Study
Arm/Group | Patients Injured
Started | 231
Completed | 231
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients evaluated at OHSU Hospital with horse related injuries
Arm/Group | Patients Injured
Number analyzed (Participants) | 231
Age, Continuous [Mean (Full Range); unit: years] | 38 [2 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 231

OUTCOME MEASURES:

1. Primary Outcome: Injury Severity Score (ISS)
Description: The Injury Severity Score (ISS) is based upon the Abbreviated Injury Scale (AIS) and is calculated by dividing the body into 6 regions. Each region is scored on a scale of 1 (minor severity/better) to 5 (most severity/worse). ISS total score is calculated by squaring each of the 3 most severely injured body regions, then summing the three squared numbers. Total ISS score can range from 3 to 75.
Time Frame: 2008-2011
Population: All patients evaluated at OHSU Hospital with horse-related injuries
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Patients Injured: All patients evaluated at OHSU Hospital with horse-related injuries
Arm/Group | Patients Injured
Number analyzed (Participants) | 231
units on a scale | 11.3 [1 to 45]

2. Other Pre Specified Outcome: Helmet Use
Description: Those patients who were wearing a helmet at the time of injury
Time Frame: 2001-2008
Measure: Number; unit: percentage of participants
Groups:
- Helmet Use: Those patients wearing a helmet at the time of injury
Arm/Group | Helmet Use
Number analyzed (Participants) | 231
percentage of participants | 20

3. Other Pre Specified Outcome: Preventable Head Injuries
Description: Percentage of potentially preventable head injuries among those patients not wearing a helmet at the time of injury
Time Frame: 2001-2008
Measure: Number; unit: percentage of participants
Groups:
- Preventable Head Injury: Those patients not wearing a helmet at the time of injury who developed a head injury
Arm/Group | Preventable Head Injury
Number analyzed (Participants) | 172
percentage of participants | 38

4. Other Pre Specified Outcome: Hospital Cost
Description: Total inpatient hospital charges, does not include outpatient costs or any non-hospital charges such as long term therapy, insurance costs, legal cost, etc.
Time Frame: 2001-2008
Measure: Mean (Full Range); unit: US Dollars
Arm/Group | Patients Injured
Number analyzed (Participants) | 231
US Dollars | 29800 [3000 to 511000]

5. Other Pre Specified Outcome: Long Term Disability
Description: Those patients who responded to a survey regarding long term disability
Time Frame: 2001-2008
Measure: Number; unit: percentage of surveyed participants
Groups:
- Long Term Disability: Those participants who responded to a survey indicating they suffered long term disability
Arm/Group | Long Term Disability
Number analyzed (Participants) | 91
percentage of surveyed participants | 59

6. Other Pre Specified Outcome: Causes of Horse Related Injuries
Description: Causes of Horse Related Injuries as related by surveyed patients to investigators
Time Frame: 2001- 2008
Measure: Number; unit: percentage of participants
Groups:
- Poor Environmental Factors: Those patients who stated that poor environmental factors led to the injury
- Poor Horse and Rider Pairing: Those patients who stated poor horse and rider pairing led to the injury
- Equipment Failure: Those patients who stated equipment failure led to the injury
Arm/Group | Poor Environmental Factors | Poor Horse and Rider Pairing | Equipment Failure
Number analyzed (Participants) | 91 | 91 | 91
percentage of participants | 40 | 30 | 9

ADVERSE EVENTS:
Time Frame: 2001-2008
Groups:
- Participants: Patients evaluated at OHSU Hospital with horse related injuries
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/231
Serious Adverse Events (participants affected / at risk) | 0/231
Other Adverse Events (participants affected / at risk) | 0/231

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No